CLINICAL TRIAL: NCT03831880
Title: A PHASE 3, RANDOMIZED, MULTICENTER, OPEN-LABEL, CROSSOVER STUDY ASSESSING SUBJECT PERCEPTION OF TREATMENT BURDEN WITH USE OF WEEKLY GROWTH HORMONE (SOMATROGON) VERSUS DAILY GROWTH HORMONE (GENOTROPIN (REGISTERED)) INJECTIONS IN CHILDREN WITH GROWTH HORMONE DEFICIENCY
Brief Title: Patient Perception of Treatment Burden in Weekly Versus Daily Growth Hormone Injections in Children With GHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C0311002; 2018-000918-38 (EudraCT Number)
Record Dates: First submitted 2018-12-21; First posted 2019-02-06 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone; somatrogon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daily to Weekly (Other): Genotropin to somatrogon
  Interventions: Drug: Genotropin; Drug: somatrogon
- Weekly to Daily (Other): somatrogon to Genotropin
  Interventions: Drug: Genotropin; Drug: somatrogon

INTERVENTIONS:
Drug: Genotropin — Genotropin (dose [mg] at time of enrollment) given subcutaneously once daily
Drug: somatrogon — 0.66 mg/kg/week given subcutaneously once weekly

SUMMARY:
This is an open label randomized 24 week crossover trial assessing the treatment burden of a weekly growth hormone injection regimen (somatrogon) compared to a daily growth hormone injection regimen (Genotropin). Approximately 90 children with growth hormone deficiency who have been stable on treatment with daily Genotropin will be enrolled.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two sequences, either 12 weeks of continued treatment with daily Genotropin followed by 12 weeks of treatment with weekly somatrogon, or 12 weeks of treatment with weekly somatrogon followed by 12 weeks of treatment with daily Genotropin. Subjects will have study visits at Baseline, Weeks 6, 12, 18, and 24. Subjects will also be followed up by phone 8 to 12 days after each treatment period begins (Week 1 and Week 13). Subjects and caregivers (as a Dyad) will complete questionnaires assessing treatment burden at baseline and at the end of each 12 week treatment period. All subjects/caregivers will receive a follow up phone call at Week 28.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3 years old and <18 years with either isolated GHD, or GH insufficiency.
2. Currently on treatment with either Genotropin Pen®, Genotropin GoQuick Pen®, HumatroPen® (United States of America [USA] only), or Omnitrope® Pen (USA only) ≥3 months and have been compliant on a stable dose (±10%) for at least 3 months prior to screening.
3. IGF I SDS < 2.
4. Subjects on hormonal replacement therapy for other hypothalamic pituitary axis (HPA) hormonal deficiencies and/or diabetes insipidus must be on an optimized and stable treatment regimen, as determined by the Investigator, for at least 3 months prior to screening.

Exclusion Criteria

1. History of leukemia, lymphoma, sarcoma or any other cancer.
2. History of radiation therapy or chemotherapy.
3. Children with psychosocial dwarfism.
4. Children born small for gestational age (SGA) - birth weight and/or birth length < 2 SDS for gestational age.
5. Other causes of short stature such as uncontrolled primary hypothyroidism and rickets.
6. Chromosomal abnormalities including Turner's syndrome, Laron syndrome, Noonan syndrome, Prader Willi syndrome, Russell Silver syndrome, short stature homeobox (SHOX) mutations/deletions or skeletal dysplasias.
7. Treatment with regularly scheduled daily or weekly injectable medications other than Genotropin® Pen, Genotropin GoQuick®, HumatroPen® (USA only), or Omnitrope® Pen (USA only).
8. Diabetes Mellitus.
9. Current treatment with Genotropin MiniQuick.
10. History of any exposure to a long acting hGH preparation.
11. Known or suspected human immunodeficiency virus (HIV) positive patient, or patient with advanced diseases such as acquired immunodeficiency syndrome (AIDS) or tuberculosis.
12. Drug, substance, or alcohol abuse.
13. Known hypersensitivity to the components of the medication.
14. Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
15. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
16. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
17. Participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation.
18. Patient and/or the parent/legal guardian are likely to be non-compliant with respect to study conduct.
19. Subject and/or the parent/legal guardian are unable to understand written and/or verbal instructions on the proper use of growth hormone injection devices.
20. Children with closed epiphyses (this determination can be based on available existing clinical data).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (18):
  - Center of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Pediatric Endocrinology, Centennial, Colorado
  - Pediatric Endocrine Associates, PC, Greenwood Village, Colorado
  - Nemours Children's Health System, Jacksonville, Florida
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Nemours Biomedical Research, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - Shriners Hospitals for Children, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - IU Health Pharmacy, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - MultiCare Health System - Mary Bridge Children's Health Center, Tacoma, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- First Pediatric Clinic UMHAT "St. Marina" EAD, Varna, Bulgaria
- Czechia (4):
  - Fakultni nemocnice Brno, Pediatricka Klinika, Brno
  - Nemocnicni lekarna FN Brno, Brno
  - Fakultni nemocnice v Motole, Pediatricka klinika 2.LF UK a FN Motol, Prague
  - Nemocnicni lekarna FN Motol, Prague
- Slovakia (4):
  - Nemocnicna Lekaren Nudch, Bratislava
  - Národný ústav detských chorôb, Detská klinika, Bratislava
  - Detská fakultná nemocnica Košice Klinika detí a dorastu LF UPJŠ a DFN, Košice
  - Nemocnica lekaren DFN Kosice, Klinika deti a dorastu, Košice
- United Kingdom (5):
  - St. Georges University Hospitals NHS Foundation Trust, London
  - St. Georges University Hospital NHS Foundation Trust, London
  - The Institute of Child Health, University College London, London
  - Great Ormond Street Hospital, London
  - NIHR Clinical Research Facility, Great Ormond Street Hospital for Children NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0311002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 107 participants were screened for study eligibility. 87 Participants, aged 3 to less than 18 years with growth hormone deficiency (GHD) on stable treatment with somatropin, were deemed eligible for enrollment and randomized to receive treatment.
Groups:
- Daily Genotropin Then Weekly Somatrogon: Participants were randomized to receive Genotropin, daily subcutaneously at the same dose which they were receiving at the time of enrollment, for 12 weeks in Period 1. Period 1 was followed by Period 2, where participants received Somatrogon, weekly subcutaneously at a dose of 0.66 milligram per kilogram per week (mg/kg/week) for 12 weeks. There was no treatment wash-out period since these participants had to take growth hormone continually. Participants were followed up maximum for 35 days (5 weeks) after last dose of study drug.
- Weekly Somatrogon Then Daily Genotropin: Participants were randomized to receive Somatrogon, weekly subcutaneously at a dose of 0.66 mg/kg/week, for 12 weeks in Period 1. Period 1 was followed by Period 2, where participants continued to receive Genotropin, daily subcutaneously at the same dose which they were receiving at the time of enrollment, for 12 weeks. There was no treatment wash-out period since these participants had to take growth hormone continually. Participants were followed up maximum for 35 days after last dose of study drug.
Period: Period 1 (12 Weeks)
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Started | 43 | 44
Completed | 43 | 43
Not Completed | 0 | 1
Not completed — Adverse event, not serious | 0 | 1
Period: Period 2 (12 Weeks)
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Started | 43 | 43
Completed | 43 | 42
Not Completed | 0 | 1
Not completed — Protocol Deviation | 0 | 1
Period: Follow-up (5 Weeks)
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Started | 43 | 43 (1 participant who discontinued from Period 1 completed follow-up visit.)
Completed | 43 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study intervention. The participants were analyzed according to the intervention they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.8 (3.4) | 10.7 (3.7) | 10.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 34 | 38 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 39 | 42 | 81
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 39 | 42 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Score Related to Overall Life Interference Assessed at Baseline, Using Dyad Clinical Outcomes Assessment 1 (DCOA 1) Questionnaire
Description: Participants were assessed for their treatment burden using DCOA 1 questionnaire completed by participant/caregiver dyads. The participant life interference questionnaire component of the DCOA 1 had 7 questions (life interference [5 questions]: a measure of life interference [daily activities/social activities/leisure/night away from home/travel]; life interference-changes to life routine [1 question]: a measure of how often changes are made to life routine; and life interference-bother of growth hormone [GH] injections [1 question]: a measure of how often the growth hormone injections cause bother) and all questions used a 5-point scale: 1= never, 2= rarely, 3= sometimes, 4= often, 5= always. The overall life interference total score was sum of all 7 questions, scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant less life interference (better outcome).
Time Frame: Baseline
Population: The full analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 40
units on a scale | 29.5 (18.0) | 27.1 (19.8)

2. Primary Outcome: Total Score Related to Overall Life Interference Assessed at Week 12, Using DCOA 1 Questionnaire
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 40
units on a scale | 25.2 (17.3) | 7.1 (7.8)

3. Primary Outcome: Total Score Related to Overall Life Interference Assessed at Week 24, Using DCOA 1 Questionnaire
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
units on a scale | 9.5 (13.3) | 23.0 (22.6)

4. Primary Outcome: Total Score Related to Overall Life Interference by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 1
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Genotropin: Participants received Genotropin, daily subcutaneously, in overall study (either in Period 1 or in Period 2).
- Somatrogon: Participants received Somatrogon, weekly subcutaneously, at a dose of 0.66 mg/kg/week, in overall study (either in Period 1 or in Period 2).
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 24.13 [20.61 to 27.65] | 8.63 [5.05 to 12.22]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p < 0.0001, Mixed Models Analysis — 95% CI: Model-based difference in means. Results were based on a linear mixed effects model including sequence, period, and treatment as fixed effects and participant within sequence and within-participant error as random effects; Mean Difference (Final Values) = -15.49, 95% CI 2-sided [-19.71 to -11.27]

5. Secondary Outcome: Total Score Related to Pen Ease of Use Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked 5 questions from Section I of the Injection Pen Assessment Questionnaire (IPAQ) patient-reported outcome (PRO) tool related to pen ease of use and used a 5-point scale: 1= very easy, 2= somewhat easy, 3= neither easy nor difficult, 4= somewhat difficult, 5= very difficult. The total score related to pen ease of use was sum of all 5 questions; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: The full analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention. Here 'number analyzed' signifies participants evaluable for each specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 10.6 (11.3) | 11.6 (12.8)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 12.0 (13.8) | 5.1 (7.6)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 5.5 (9.3) | 9.4 (13.0)

6. Secondary Outcome: Total Score Related to Pen Ease of Use by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked 5 questions from Section I of the IPAQ PRO tool related to pen ease of use and used a 5-point scale: 1= very easy, 2= somewhat easy, 3= neither easy nor difficult, 4= somewhat difficult, 5= very difficult. The total score related to pen ease of use was sum of all 5 questions; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant a better outcome.
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 10.71 [8.27 to 13.14] | 5.32 [2.84 to 7.80]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p = 0.0017, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -5.39, 95% CI 2-sided [-8.69 to -2.09]

7. Secondary Outcome: Total Score Related to Ease of the Injection Schedule Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked a question from Section I of the IPAQ PRO tool related to ease of injection schedule and used a 5-point scale: 1= very easy, 2= somewhat easy, 3= neither easy nor difficult, 4= somewhat difficult, 5= very difficult. The total score related to ease of the injection schedule ranged from 1 to 5; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 18.5 (20.0) | 16.3 (17.5)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 23.3 (25.2) | 4.4 (11.2)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 9.5 (18.3) | 17.9 (22.3)

8. Secondary Outcome: Total Score Related to Ease of the Injection Schedule by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 7
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 20.56 [16.22 to 24.89] | 6.96 [2.54 to 11.37]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -13.60, 95% CI 2-sided [-19.74 to -7.45]

9. Secondary Outcome: Total Score Related to Convenience of the Injection Schedule Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked a question from Section I of the IPAQ PRO tool related to ease of injection schedule and used a 7-point scale: 1=extremely convenient to 7=extremely inconvenient. The total score related to convenience of injection schedule ranged from 1 to 7; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 34.5 (21.0) | 32.5 (21.3)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 35.3 (23.9) | 7.9 (10.7)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 11.9 (14.4) | 33.3 (24.1)

10. Secondary Outcome: Total Score Related to Convenience of the Injection Schedule by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 9
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 34.30 [30.13 to 38.47] | 9.96 [5.71 to 14.21]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -24.34, 95% CI 2-sided [-30.10 to -18.57]

11. Secondary Outcome: Total Score Related to Satisfaction With Overall Treatment Experience Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked a question from Section I of the IPAQ PRO tool related to participant satisfaction with treatment and used a 5-point scale: 1=very satisfied to 5=very dissatisfied. The total score related to satisfaction with overall treatment ranged from 1 to 5; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 28.0 (21.5) | 29.4 (23.3)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 27.3 (27.2) | 20.0 (31.1)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 22.0 (32.3) | 30.4 (27.9)

12. Secondary Outcome: Total Score Related to Satisfaction With Overall Treatment Experience by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 11
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 28.95 [22.55 to 35.36] | 21.13 [14.61 to 27.65]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p = 0.0739, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -7.83, 95% CI 2-sided [-16.42 to 0.77]

13. Secondary Outcome: Total Scores Related to Willingness to Continue Injection Schedule Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked a question from Section I of the IPAQ PRO tool related to participant willingness to continue treatment and used a 5-point scale: 1=extremely willing to 5=not at all willing. The total score related to willingness to continue injection schedule ranged from 1 to 5; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 42 | 40
  Baseline | 18.5 (20.0) | 22.5 (23.9)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 28.5 (27.6) | 10.6 (21.1)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 13.1 (24.8) | 30.4 (29.0)

14. Secondary Outcome: Total Scores Related to Willingness to Continue Injection Schedule by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 13
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 29.54 [23.95 to 35.12] | 11.93 [6.24 to 17.62]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -17.60, 95% CI 2-sided [-25.15 to -10.06]

15. Secondary Outcome: Total Scores Related to Injection Signs and Symptoms for Participants Aged 8 Years and Above Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participants (8-17 years old). Participants were asked 4 questions from Section I of the IPAQ PRO tool related to participant's injection signs and symptoms and used a 11-point scale: 0=no pain to 10=worst possible pain; 0=no stinging to 10=worst possible stinging; 0=no bruising to 10=worst possible bruising; and 0=no bleeding to 10=worst possible bleeding, respectively. The total score was sum of all questions; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score for injection signs and symptoms meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: The full analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Here 'number analyzed' signifies participants aged 8 years or above and evaluable for each specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 35 | 34
units on a scale
  Baseline: number analyzed (Participants) | 35 | 29
  Baseline | 15.0 (10.4) | 13.8 (11.9)
  Week 12: number analyzed (Participants) | 34 | 25
  Week 12 | 16.2 (12.2) | 13.7 (10.3)
  Week 24: number analyzed (Participants) | 32 | 32
  Week 24 | 13.6 (12.2) | 10.9 (9.6)

16. Secondary Outcome: Total Scores Related to Injection Signs and Symptoms for Participants Aged 8 Years and Above by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 15
Time Frame: Baseline up to Week 24
Population: The full analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention. Here "Overall number of participants analyzed" signifies participants aged 8 years or above and evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 66 | 57
units on a scale | 13.56 [10.78 to 16.34] | 14.27 [11.32 to 17.21]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p = 0.6137, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-2.09 to 3.51]

17. Secondary Outcome: Total Scores Related to Assessment of Signs, Completed by Caregiver for Children Aged <8 Years Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by caregiver for children under 8 years. Participants were asked 2 questions from Section I of the IPAQ PRO tool related to participant's assessment of signs and used a 11-point scale: 0=no bruising to 10=worst possible bruising and 0=no bleeding to 10=worst possible bleeding, respectively. The total score was sum of all questions; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score for assessment of signs meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: The full analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure. Here 'number analyzed' signifies participants aged 8 years or below and evaluable for each specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 8 | 10
units on a scale
  Baseline: number analyzed (Participants) | 6 | 10
  Baseline | 14.2 (14.6) | 13.5 (11.3)
  Week 12: number analyzed (Participants) | 7 | 10
  Week 12 | 9.3 (10.6) | 13.0 (15.8)
  Week 24: number analyzed (Participants) | 8 | 9
  Week 24 | 5.6 (7.8) | 9.4 (8.8)

18. Secondary Outcome: Total Scores Related to Assessment of Signs, Completed by Caregiver for Children Aged <8 Years by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 17
Time Frame: Baseline up to Week 24
Population: The full analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention. Here "Overall number of participants analyzed" signifies participants aged 8 years or below and evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 16 | 18
units on a scale | 8.75 [2.65 to 14.86] | 9.31 [3.47 to 15.16]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p = 0.8404, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-5.29 to 6.41]

19. Secondary Outcome: Total Scores Related to Caregiver Life Interference, Including Family Life Interference Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by caregiver. Participants were asked 13 questions from Section I of the IPAQ PRO tool related to caregiver life interference and used a 5-point scale: 1= never to 5= always. The total score ranged was sum of scores from all questions; scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score for caregiver and family life interference meant less life interference (a better outcome).
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 41 | 40
  Baseline | 17.8 (17.5) | 20.0 (20.1)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 15.9 (16.7) | 3.1 (5.5)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 3.8 (6.0) | 18.1 (23.4)

20. Secondary Outcome: Total Scores Related to Caregiver Life Interference, Including Family Life Interference by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 19
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 17.01 [13.77 to 20.25] | 3.54 [0.24 to 6.84]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -13.47, 95% CI 2-sided [-17.59 to -9.35]

21. Secondary Outcome: Total Scores Related to Missed Injections Assessed at Baseline, Week 12 and Week 24, Using DCOA 1 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 1 questionnaire completed by participant/caregiver dyads. Participants were asked a question from Section I of the IPAQ PRO tool related to number of missed injections (daily or weekly administration) during past 4 weeks. The total scores ranged from 0 to 31 for daily administration (Genotropin) and from 0 to 5 for weekly administration (Somatrogon). All scores were transformed from raw scores and converted to a 0 to 100 scale; a lower score for missed injections meant a better outcome.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 41 | 40
  Baseline | 7.8 (15.1) | 7.3 (16.1)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 4.3 (8.2) | 0.0 (0.0)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 1.9 (7.4) | 3.1 (10.8)

22. Secondary Outcome: Total Scores Related to Missed Injections by Treatment in Overall Study, Using DCOA 1 Questionnaire
Description: as for outcome 21
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 3.71 [2.03 to 5.39] | 0.95 [-0.76 to 2.66]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p = 0.0245, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.76, 95% CI 2-sided [-5.16 to -0.36]

23. Secondary Outcome: Number of Participants as Per Responses to Choice of Injection Pen Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregivers responded to question from Section II of the IPAQ PRO tool "If you were given the choice between the daily growth hormone injection pen and the weekly growth hormone injection pen, which pen would you choose?" Response was: 1) the daily injection pen (Genotropin) or 2) the weekly injection pen (Somatrogon).
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Somatrogon | 38 | 36
  Genotropin | 4 | 6

24. Secondary Outcome: Number of Participants as Per Responses to Preferred Injection Schedule Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregivers responded to question from Section II of the IPAQ PRO tool "Which growth hormone injection schedule do you prefer overall?" by choosing from any 1 option from: 1) prefer the weekly injection schedule (Somatrogon); 2) prefer the daily injection schedule (Genotropin); 3) no preference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Somatrogon | 40 | 37
  Genotropin | 2 | 4
  No Preference | 0 | 1

25. Secondary Outcome: Number of Participants as Per Responses to Convenience of the Injection Schedule Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregivers responded to question from Section II of the IPAQ PRO tool "Which growth hormone injection schedule was more convenient overall?" by choosing from any 1 option from: 1) weekly injection schedule was more convenient (Somatrogon); 2) daily injection schedule was more convenient (Genotropin); 3) no difference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Somatrogon | 40 | 40
  Genotropin | 2 | 2
  No Difference | 0 | 0

26. Secondary Outcome: Number of Participants as Per Responses to Ease of Following Injection Schedule Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregivers responded to question from Section II of the IPAQ PRO tool "Which growth hormone injection schedule was easier to follow overall?" by choosing from any 1 option from: 1) easier to follow weekly injection schedule (Somatrogon); 2) easier to follow daily injection schedule (Genotropin); 3) no difference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Somatrogon | 38 | 34
  Genotropin | 4 | 4
  No Difference | 0 | 4

27. Secondary Outcome: Number of Participants as Per Responses to Pen Ease of Use Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregiver were asked a question "Which pen was easier to use?" from Section II of the IPAQ PRO tool. Question had 4 parts: preparing the injection pen (Part I), setting the dose (Part II), injecting the medicine (Part III) and storing the pen (Part IV). Participants/caregiver expressed their preference by choosing from any 1 option for each activity from: 1) weekly pen easier to use (Somatrogon); 2) daily pen easier to use (Genotropin); 3) no difference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Part I: Somatrogon | 29 | 25
  Part I: Genotropin | 3 | 4
  Part I: No difference | 10 | 13
  Part II: Somatrogon | 21 | 17
  Part II: Genotropin | 6 | 8
  Part II: No Difference | 15 | 17
  Part III: Somatrogon | 13 | 18
  Part III: Genotropin | 16 | 12
  Part III: No Difference | 13 | 12
  Part IV: Somatrogon | 12 | 14
  Part IV: Genotropin | 2 | 2
  Part IV: No Difference | 28 | 26

28. Secondary Outcome: Number of Participants as Per Responses to Participant Life Interference Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregiver were asked a question "Which injection schedule interfered less?" from Section II of the IPAQ PRO tool related to participant life interference. Participants were assessed for 5 activities: daily activities (Activity 1), social activities (Activity 2), recreation/leisure activities (Activity 3), spending night away from home (Activity 4) and travel (Activity 5). The participants expressed their preference by choosing from any 1 option for each activity from: 1) weekly injection schedule interfered less (Somatrogon); 2) daily injection schedule interfered less (Genotropin); 3) no difference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Activity 1: Somatrogon | 35 | 31
  Activity 1: Genotropin | 2 | 1
  Activity 1: No Difference | 5 | 10
  Activity 2: Somatrogon | 34 | 34
  Activity 2: Genotropin | 2 | 0
  Activity 2: No Difference | 6 | 8
  Activity 3: Somatrogon | 34 | 33
  Activity 3: Genotropin | 2 | 1
  Activity 3: No Difference | 6 | 8
  Activity 4: Somatrogon | 36 | 37
  Activity 4: Genotropin | 2 | 1
  Activity 4: No Difference | 4 | 4
  Activity 5: Somatrogon | 33 | 37
  Activity 5: Genotropin | 3 | 0
  Activity 5: No Difference | 6 | 5

29. Secondary Outcome: Number of Participants as Per Responses to Caregiver Life Interference Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Caregivers of participants were asked a question "Which injection schedule interfered less?" from Section II of the IPAQ PRO tool related to caregiver life interference and were assessed for 5 activities: daily activities (Activity 1), social activities (Activity 2), recreation/leisure activities (Activity 3), spending night away from home (Activity 4) and travel (Activity 5). Preference was expressed by choosing from any 1 option for each activity from: 1) weekly injection schedule interfered less (Somatrogon); 2) daily injection schedule interfered less (Genotropin); 3) no difference. The caregivers responded for the participants, and in actual they respond to the number of participants only but per caregiver responses.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Activity 1: Somatrogon | 36 | 31
  Activity 1: Genotropin | 2 | 0
  Activity 1: No Difference | 4 | 11
  Activity 2: Somatrogon | 36 | 32
  Activity 2: Genotropin | 2 | 0
  Activity 2: No Difference | 4 | 10
  Activity 3: Somatrogon | 35 | 34
  Activity 3: Genotropin | 2 | 0
  Activity 3: No Difference | 5 | 8
  Activity 4: Somatrogon | 35 | 37
  Activity 4: Genotropin | 1 | 0
  Activity 4: No Difference | 6 | 5
  Activity 5: Somatrogon | 35 | 37
  Activity 5: Genotropin | 2 | 0
  Activity 5: No Difference | 5 | 5

30. Secondary Outcome: Number of Participants as Per Responses to Family Life Interference Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/ caregiver were asked a question "Which injection schedule interfered less?" from Section II of the IPAQ PRO tool related to family life interference and assessed for 5 activities: daily activities (Activity 1), social activities (Activity 2), recreation/leisure activities (Activity 3), spending night away from home (Activity 4) and travel (Activity 5). Preference was expressed by choosing from any 1 option for each activity from: 1) weekly injection schedule interfered less (Somatrogon); 2) daily injection schedule interfered less (Genotropin); 3) no difference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Activity 1: Somatrogon | 32 | 29
  Activity 1: Genotropin | 1 | 0
  Activity 1: No Difference | 9 | 13
  Activity 2: Somatrogon | 32 | 30
  Activity 2: Genotropin | 1 | 0
  Activity 2: No Difference | 9 | 12
  Activity 3: Somatrogon | 32 | 32
  Activity 3: Genotropin | 1 | 0
  Activity 3: No Difference | 9 | 10
  Activity 4: Somatrogon | 31 | 34
  Activity 4: Genotropin | 1 | 0
  Activity 4: No Difference | 10 | 8
  Activity 5: Somatrogon | 31 | 36
  Activity 5: Genotropin | 1 | 0
  Activity 5: No Difference | 10 | 6

31. Secondary Outcome: Number of Participants as Per Response to Benefit Relating to the Injection Schedule Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants were assessed for their treatment experience using DCOA 2 questionnaire completed by participant/caregiver dyads. Participants/caregiver were asked a question "How beneficial was to take injections less often?" from Section II of the IPAQ PRO tool pertaining to benefit relating to the Injection schedule and used a 5-point scale: 1= extremely beneficial, 2= very beneficial, 3= moderately beneficial, 4= slightly beneficial and 5= not at all beneficial. Lower score of benefit relating to injection schedule meant a better outcome.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Extremely Beneficial | 28 | 20
  Very Beneficial | 11 | 14
  Moderately Beneficial | 1 | 3
  Slightly Beneficial | 0 | 3
  Not At All Beneficial | 2 | 2

32. Secondary Outcome: Number of Participants as Per Responses to Intention to Comply Assessed at Week 24, Using DCOA 2 Questionnaire
Description: Participants/caregiver dyads were asked 4 questions "Which schedule would be better able to follow?" (Question 1), "Which schedule would be more likely to follow for a longer time?" (Question 2), "Which schedule would be better able to follow for a longer time?" (Question 3) and "Which schedule would be more likely to follow?" (Question 4) from Section II of the IPAQ PRO tool related to participant intention to comply with treatment. Options for each question were: 1) weekly injection (Somatrogon) 2) daily injection (Genotropin), or 3) no difference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 42 | 42
Participants
  Question 1: Somatrogon | 33 | 31
  Question 1: Genotropin | 2 | 2
  Question 1: No Difference | 7 | 9
  Question 2: Somatrogon | 29 | 32
  Question 2: Genotropin | 1 | 2
  Question 2: No Difference | 12 | 8
  Question 3: Somatrogon | 34 | 35
  Question 3: Genotropin | 1 | 1
  Question 3: No Difference | 7 | 6
  Question 4: Somatrogon | 26 | 31
  Question 4: Genotropin | 3 | 2
  Question 4: No Difference | 13 | 9

33. Secondary Outcome: Patient Global Impression Severity-Impact on Daily Activities (PGIS-IDA) Score Assessed at Baseline, Week 12 and Week 24
Description: The PGIS-IDA rated the severity of the impact on daily activities due to the treatment administration during the past 4 weeks on a 7-point scale (1= not present to 7= extremely severe). Scores were transformed from raw scores to a 0 to 100 scale. Lower scores meant less impact on daily activities (better outcome).
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
units on a scale
  Baseline: number analyzed (Participants) | 41 | 40
  Baseline | 15.0 (14.8) | 16.3 (16.2)
  Week 12: number analyzed (Participants) | 43 | 40
  Week 12 | 19.0 (19.4) | 4.6 (7.5)
  Week 24: number analyzed (Participants) | 42 | 42
  Week 24 | 7.1 (9.8) | 22.2 (20.4)

34. Secondary Outcome: Patient Global Impression Severity-Impact on Daily Activities (PGIS-IDA) Score by Treatment in Overall Study
Description: as for outcome 33
Time Frame: Baseline up to Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 85 | 82
units on a scale | 20.64 [17.30 to 23.99] | 6.06 [2.66 to 9.46]
Statistical Analysis 1: Comparison: Genotropin vs Somatrogon; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -14.58, 95% CI 2-sided [-18.72 to -10.44]

35. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Emergent Treatment Related AEs and SAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Treatment-emergent AEs (TEAEs) were defined as events that occurred between first dose of study drug up to 35 days after last dose of study drug. Related TEAEs were those AEs who had relation to the study treatment and was judged by investigator.
Time Frame: Baseline up to 35 days after last dose of study drug (up to 29 Weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 86 | 87
Participants
  Treatment-Emergent AEs | 38 | 47
  Treatment-Emergent SAEs | 0 | 0
  Treatment-Emergent Related AEs | 14 | 21
  Treatment-Emergent Related SAEs | 0 | 0

36. Other Pre Specified Outcome: Number of Participants With Adverse Events According to Severity
Description: AEs were assessed and categorized according to the severity as mild (did not interfered with participant's usual function), moderate (interfered to some extent with participant's usual function) and severe (interfered significantly with participant's usual function).
Time Frame: Baseline up to 35 days after last dose of study drug (up to 29 Weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 86 | 87
Participants
  Mild | 34 | 41
  Moderate | 4 | 6
  Severe | 0 | 0

37. Other Pre Specified Outcome: Number of Participants With Discontinuation Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The discontinuations due to adverse events was defined for participants and reported in this outcome measure.
Time Frame: Baseline up to 35 days after last dose of study drug (up to 29 Weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Genotropin | Somatrogon
Number analyzed (Participants) | 86 | 87
Participants | 0 | 1

38. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: The laboratory abnormality parameters included Hematology: erythrocyte (Er.) mean corpuscular volume, Er. mean corpuscular hemoglobin:<0.9*lower limit normal (LLN), leukocytes:<0.6*LLN, lymphocytes:<0.8*LLN, neutrophils:<0.8*LLN, greater than (>) 1.2*upper limit normal (ULN), eosinophils, monocytes:>1.2*ULN. Clinical chemistry: bilirubin, direct bilirubin, indirect bilirubin:>1.5*ULN, gamma glutamyl transferase:>3.0*ULN, albumin:>1.2*ULN, blood urea nitrogen:>1.3*ULN, urate:>1.2*ULN, high-density lipoprotein (HDL) cholesterol:<0.8*LLN, potassium, magnesium:>1.1*ULN, phosphate:>1.2*ULN, bicarbonate:<0.9*LLN, creatine kinase:>2.0*ULN. Urinalysis: specific gravity:>1.030, ketones, urine protein, urine hemoglobin, nitrite, leukocyte esterase:>=1.
Time Frame: Week 1 to Week 12, Week 13 to Week 24
Population: The safety analysis set included all participants who received at least 1 dose of study intervention. The participants were analyzed according to the intervention they actually received. Here 'number analyzed' signifies participants evaluable for each specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
Participants
  Week 1 to Week 12: number analyzed (Participants) | 41 | 36
  Week 1 to Week 12 | 19 | 19
  Week 13 to Week 24: number analyzed (Participants) | 42 | 43
  Week 13 to Week 24 | 24 | 21

39. Other Pre Specified Outcome: Number of Participants With Positive Anti-Recombinant Human Growth Hormone (rhGH) Antibodies and Neutralizing Antibodies (NAb)
Description: Blood samples were collected for determination of rhGH and NAb. The participants who tested positive for antibodies were reported.
Time Frame: Baseline, Week 12, Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
Participants
  Baseline: Anti-rhGH | 5 | 0
  Baseline: Neutralizing | 0 | 0
  Week 12: Anti-rhGH | 3 | 3
  Week 12: Neutralizing | 0 | 0
  Week 24: Anti-rhGH | 4 | 6
  Week 24: Neutralizing | 0 | 0

40. Other Pre Specified Outcome: Number of Participants With Positive Anti-Somatrogon Antibodies and Neutralizing Antibodies (NAb)
Description: Blood samples were collected for determination of anti-somatrogon antibodies and NAb. The participants who tested positive for antibodies were reported.
Time Frame: Baseline, Week 12, Week 24
Population: The safety analysis set included all participants who received at least 1 dose of study intervention. The participants were analyzed according to the intervention they actually received. "0" in number analyzed field denotes that participants who followed the 'Genotropin then Somatrogon' sequence were not tested for anti-somatrogon ADA at Week 12 and participants who followed the 'Somatrogon then Genotropin' sequence were not tested for anti-somatrogon ADA at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Genotropin Then Weekly Somatrogon | Weekly Somatrogon Then Daily Genotropin
Number analyzed (Participants) | 43 | 44
Participants
  Baseline: Anti-Somatrogon Antibodies | 0 | 0
  Baseline: Neutralizing | 0 | 0
  Week 12: Anti-Somatrogon Antibodies: number analyzed (Participants) | 0 | 44
  Week 12: Anti-Somatrogon Antibodies |  | 4
  Week 12: Neutralizing: number analyzed (Participants) | 0 | 44
  Week 12: Neutralizing |  | 0
  Week 24: Anti-Somatrogon Antibodies: number analyzed (Participants) | 43 | 0
  Week 24: Anti-Somatrogon Antibodies | 0 |
  Week 24: Neutralizing: number analyzed (Participants) | 43 | 0
  Week 24: Neutralizing | 0 |

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days after last dose of study drug (up to 29 weeks)
Description: Adverse events reported here are per treatment participants received during the study (either in Period 1 or Period 2). Safety set was evaluated.
Arm/Group | Genotropin | Somatrogon
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 38/86 | 47/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin (N=86) | Somatrogon (N=87)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Administration site oedema (General disorders) | 0 | 1
Administration site pain (General disorders) | 0 | 2
Application site pruritus (General disorders) | 1 | 0
Fat tissue increased (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Injection site bruising (General disorders) | 2 | 1
Injection site erythema (General disorders) | 1 | 1
Injection site haematoma (General disorders) | 8 | 4
Injection site haemorrhage (General disorders) | 2 | 0
Injection site pain (General disorders) | 11 | 13
Injection site reaction (General disorders) | 0 | 1
Injection site swelling (General disorders) | 2 | 2
Pyrexia (General disorders) | 4 | 2
Hypersensitivity (Immune system disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 6
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 3 | 1
Viral rash (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Body temperature increased (Investigations) | 1 | 3
Insulin-like growth factor increased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 6
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Excessive exercise (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03831880/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03831880/SAP_001.pdf